CLINICAL TRIAL: NCT03915574
Title: Dural Puncture Epidural Versus Epidural Anesthesia for Cesarean Delivery: A Randomized, Double-blind Study
Brief Title: Dural Puncture Epidural Versus Epidural Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 228768
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-10

CONDITIONS: Pain Levels

STUDY DESIGN:
Intervention Model Description: 140 mother-infant dyads (280 actual participants)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dural Puncture Epidural (Experimental): Participants will receive a dural puncture epidural block with a 25 gauge spinal needle followed by a standard epidural infusion (0.0625% bupivacaine + 2mcg/ml fentanyl)
  Interventions: Device: 25G Dural Puncture Epidural
- Standard Epidural (Active Comparator): Participants will have standard epidural infusion followed by a standard epidural infusion (0.0625% bupivacaine + 2mcg/ml fentanyl)
  Interventions: Device: Standard Epidural

INTERVENTIONS:
Device: 25G Dural Puncture Epidural — Dural puncture created with a 25 gauge spinal needle
  Arms: Dural Puncture Epidural
Device: Standard Epidural — Control group - standard epidural (no dural puncture)
  Arms: Standard Epidural

SUMMARY:
This study will compare two anesthetics techniques called Dural Puncture Epidural (DPE) and Standard Epidural as to which of the two can provide faster and potentially better at providing pain relief for cesarean sections. It will also compare these two anesthetics techniques on the percentage of women who require additional drugs to control pain during their cesarean deliveries. The results of this study will help anesthesiologists know which anesthetic technique can provide faster and potentially better at providing pain relief for cesarean sections.

DETAILED DESCRIPTION:
The aim of this study is to compare the onset time of anesthesia between standard epidural and Dural Puncture Epidural (DPE) for cesarean delivery. The study will hypothesize that a DPE technique with a 25-gauge spinal needle will have a faster onset and improved quality of surgical anesthesia when compared to a standard epidural. Participants will be blinded to which group they are being assigned. An unblinded anesthesiologist will insert the epidural or DPE based on randomization. After insertion of the epidural or DPE, a low dose local anesthetic infusion will be infused into the epidural catheter up until the time of surgery. This is the standard infusion used to provide pain relief in laboring women (bupivacaine 0.0625% with 2 mcg/ml fentanyl). In this way participants enrolled in the study would mimic anesthetic the conditions of a "labor epidural".

Participants will then move on to the next phase of the study. In this phase, the epidural pump will be discontinued, and anesthesia care will be conducted in the same manner as all cesarean deliveries under epidural extension anesthesia (this refers to the process of providing anesthesia using a pre-existing epidural/DPE that was inserted for the purpose of providing labor analgesia). Anesthesia will be induced in a standardized manner with 20 ml of 3% chloroprocaine. Motor and sensory block will be tested at the end of the epidural loading dose. Loss of sharp sensation will be measured using a blunt plastic neurotip® (Owen Mumford, USA) until a sensory bilateral block to the T6 dermatomal level has been reached. The T6 level measured at the xiphoid process will be marked bilaterally with a washable marker pen to guarantee the precision of the primary endpoint (which will be assumed when sensory block goes above T6). Sensory testing will be performed from caudad to cephalad (i.e. from blocked to unblocked dermatomes) to identify the first unblocked dermatome. To identify the level where the sensation of touch is first appreciated, the investigator will ask the question: "Tell me when you feel the sensation of something sharp touching your skin." Both the motor and sensory block evaluations are part of the standard clinical care of patients receiving neuraxial anesthesia. The main difference for participants enrolled in the study is that the frequency of sensory assessments will be increased so that the onset of surgical anesthesia can be accurately documented (approximately every minute and then more frequently as the sensory block approaches the primary endpoints). A second anesthesiologist, blind to the type of block will manage the clinical care of the patient from the beginning of the study (after epidural catheter placement) and will administer the induction drug (prepared by that anesthesiologist as per SOC). There will be no difference in this clinician's care of the subject than if she were not enrolled in the study. This will assess the onset of anesthesia and manage all aspects of the subject's clinical care including the documentation of the local anesthetic (LA) solution administration timing and its clinical effects. The speed of onset will be assessed from the end of epidural test dose. This will be defined as time zero and the start of anesthesia. If required, intra-operative analgesia will be offered in the form of further epidural top-up, intravenous fentanyl, ketamine, nitrous oxide or replacement of neuraxial anesthesia/conversion into general anesthesia as the standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestation > 36 weeks
* ASA class II and III
* Provides written consent
* Infant of mother
* Elective or non-urgent cesarean delivery

Exclusion Criteria:

* Patient refusal
* Urgent/emergent cesarean sections
* ASA and IV or above
* Unable to understand English
* Significant back surgery or scoliosis
* Lethal fetal abnormality or likely to affect APGAR scores
* Weight > 120 kg
* Height < 150 cm
* Allergy to study solutions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Sharawi, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Sharawi N, Williams M, Athar W, Martinello C, Stoner K, Taylor C, Guo N, Sultan P, Mhyre JM. Effect of Dural-Puncture Epidural vs Standard Epidural for Epidural Extension on Onset Time of Surgical Anesthesia in Elective Cesarean Delivery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2326710. doi: 10.1001/jamanetworkopen.2023.26710. PMID 37526934

RESULTS

PARTICIPANT FLOW:
Groups:
- Dural Puncture Epidural: Participants will receive a dural puncture epidural block with a 25 gauge spinal needle and a loading dose of 10 - 20 ml of 0.0625% bupivacaine + 2mcg/ml fentanyl, followed by an epidural infusion of the same medications
  25G Dural Puncture Epidural: Dural puncture created with a 25 gauge spinal needle
- Standard Epidural: Participants will receive a standard epidural and a loading dose of 10 - 20 ml of 0.0625% bupivacaine + 2mcg/ml fentanyl, followed by an epidural infusion of the same medications
  Standard Epidural: Control group - standard epidural (no dural puncture)
Period: Overall Study
Arm/Group | Dural Puncture Epidural | Standard Epidural
Started | 70 (70 mother-infant dyads (total participants = 140 per arm)) | 70 (70 mother-infant dyads (total participants = 140 per arm))
Completed | 70 (70 mother-infant dyads completed the study (total participants = 140)) | 66 (66 mother-infant dyads completed the study (participants = 132))
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: 70 mother-infant dyads per arm, Baseline characteristics not collected for infants, Infants were not monitored for adverse events
Groups:
- Total: Total of all reporting groups
Arm/Group | Dural Puncture Epidural | Standard Epidural | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.3) | 31 (5.1) | 30.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 4 participants in the Standard Epidural Arm did not receive the allocated intervention, so Race data was not collected for 4 participants
  Participants
    number analyzed (Participants) | 70 | 66 | 136
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 27 | 19 | 46
    White | 40 | 45 | 85
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 3 | 0 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index is calculated as weight in kilograms divided by height in meters squared
  kg/m^2 | 33.9 (6.4) | 32.9 (4.9) | 33.4 (5.65)

OUTCOME MEASURES:

1. Primary Outcome: Onset Time of Surgical Anesthesia
Description: The primary outcome will be the onset time of surgical anesthesia in seconds. This will be measured from the induction of anesthesia (as defined by the beginning of injection of the "Induction 1 syringe") to the point at which sharp sensation is lost bilaterally at the T6 dermatomal level (as measured by a blunt plastic neurotip® (Owen Mumford, USA) device)
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Dural Puncture Epidural | Standard Epidural
Number analyzed (Participants) | 70 | 66
seconds | 422 [290 to 546] | 655 [437 to 926]

2. Secondary Outcome: Number of Participants With Inadequate Neuraxial Analgesia or Anesthesia
Description: A composite outcome defined by failure to achieve at least a T10 bilateral sensory level pre-operatively (after 3 ml 1.5% lidocaine with 1:200,000 epinephrine 45 mg lidocaine and up to 20 ml of 0.0625% bupivacaine with 2mcg/ml fentanyl), the requirement for intraoperative analgesia supplementation, conversion to general anesthesia or repeat neuraxial procedure, or failure to achieve the primary outcome within 15 minutes between the two groups. Analyzed as a collapsed composite (any or none)
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dural Puncture Epidural | Standard Epidural
Number analyzed (Participants) | 70 | 66
Participants | 11 | 24

3. Other Pre Specified Outcome: Maximum Pain During Surgery (Score)
Description: Maximum pain visual analogue scale during surgery (units on a scale, 0 - 10)
Time Frame: 2 hours
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Cumulative Dose of Phenylephrine Measured in Milligram Required During Surgery
Description: Vasopressor requirements during surgery required to maintain systolic blood pressure within 15% of baseline
Time Frame: 2 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patient Satisfaction With Anesthetic Technique (Score)
Description: Overall patient satisfaction score (units on a scale, 0 - 10)
Time Frame: 4 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Neonatal Requirement for Resuscitation
Description: Neonatal Apgar scores (units on a scale, 0 - 10)
Time Frame: 2 hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Neonatal Physiological Condition
Description: Umbilical cord blood gases (pH measurement)
Time Frame: 2 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Requirement for Opioids in the First 24 Hours After Surgery
Description: Opioid consumption measured in milligrams.
Time Frame: 24 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Anesthesia Side Effects
Description: nausea, vomiting, itching (yes/no)
Time Frame: 2 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Vasopressor Requirements During Surgery
Description: measured in milligrams
Time Frame: 2 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Bromage Score (0 - 3 Scale)
Description: Motor block assessment 0 - Able to move hip, knee, and ankle
  1. - unable to move hip, but able to move knee and ankle
  2. - unable to move hip and knee, but able to move ankle
  3. - unable to move hip, knee and ankle
Time Frame: 3 hours
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Sensory Block Assessment
Description: Assessed using sharp sensation at the midclavicular line on the abdomen and thorax Reported at the dermatomal level where sharp sensation is first felt
Time Frame: 3 hours
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Anesthesia Adverse Effects
Description: Accidental dural puncture, local anesthesia systemic toxicity, high spinal, post dural puncture headache
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 days
Description: Infants were not monitored for adverse events
Arm/Group | Dural Puncture Epidural | Standard Epidural
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/66
Other Adverse Events (participants affected / at risk) | 0/70 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03915574/Prot_SAP_001.pdf